CLINICAL TRIAL: NCT01022983
Title: Preoperative Levosimendan in Patients With Heart Failure Undergoing Elective Noncardiac Surgery: A Randomized, Placebocontrolled Trial. SIMPLE Study
Brief Title: Preoperative Levosimendan and Heart Failure
Acronym: PELS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Not finding patients for including
Sponsor: Sykehuset i Vestfold HF (Other)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Principal Investigator, Espen Lindholm, Seksjonsoverlege, Sykehuset i Vestfold HF
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIMPLE
Record Dates: First submitted 2009-11-24; First posted 2009-12-01 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Heart Failure; Hip Fracture
MeSH Terms: conditions — Heart Failure; Hip Fractures | interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levosimendan (Active Comparator)
  Interventions: Drug: Levosimendan
- Povidon, waterfree etanol, glucosis 5% (Placebo Comparator)
  Interventions: Drug: Levosimendan; Drug: Placebo

INTERVENTIONS:
Drug: Levosimendan — At least 2 hours before surgery: Infusion of Levosimendan (0,1 microgram/kg/min.). 24 hours of infusion without a bolus.
  Other Names: Simdax; ATC-nr.: C01C X08
Drug: Placebo — ml/kg/hours - same infusion rate as active comparator
  Arms: Povidon, waterfree etanol, glucosis 5%

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of Levosimendan given preoperative to patients with heart failure undergoing noncardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Acute surgery. Hip Fracture
* Patient with cardiac failure (EF < 35%) or known coronary disease
* At least 2 of 11 comorbidities
* Patient has to use at least one heart failure medication
* Symptoms of heart failure
* NT-proBNP > 2000pg/ml

Exclusion Criteria:

* < 18 years old
* Participants in other pharmacological study
* Abuse of medicaments or alcohol
* Pregnant or breastfeeding women
* AMI at admission
* HOCM
* Serious aortic stenosis (< 1 cm2)
* Sustained ventricular tachycardia
* Earlier episodes of "torsades de pointes"
* Sustained heartbeat > 120/minute
* Systolic BP < 90 mmHg
* Surgery planned not before 2 hours of study medication can be infused preoperative
* Cardiac surgery
* Dementia
* S-K < 3 mmol/l
* Allergy levosimendan
* Serious liver failure (Known Class C Child-Pugh score)
* Serious kidney failure (GFR < 30 ml/min.)
* Prolonged QTc-interval (male QTc > 0,43 s, female QTc > 0,45 s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Heartfailure - Highest NT-proBNP-value the first 7 days after surgery | NT-proBNP 6 hours postoperative, 24 hours postoperative, 48 h postoperative, 72 h postoperative, 96 h postoperative, 120 h postoperative, 144 h postoperative and 168 h postoperative

SECONDARY OUTCOMES:
Days of hospitalization | Hospital stay - number of days patients are hospitalized
Use of inotropes (dopamine, Norepinephrine)during postoperative unit stay. Mg/microgram | After 16-18 hours, after 48 hours and every 24 hours if still in the PO-Unit
Mortality | 30 days
  Visits or patients record
Ischemia | 7 days postoperative
  Continous ECG first 24 hours an ECG every second day
Myocardial necrosis | 7 days postoperative
  Troponin taken every day postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Espen Lindholm, MD, Study Director — Vestfold Hospital trust, Norway; Knut A Kirkebøen, PhD, Principal Investigator — Oslo University Hospital - Ullevål, Norway; Mathias Kotyra, Md, Principal Investigator — Mölndal hospital, Sweden; Anders Nydahl, Phd, Principal Investigator — University Hospital Örebro, Sweden
Locations (4):
- Norway (2):
  - Oslo University Hospital - Ullevål, Oslo
  - Vestfold Hospital Trust, Tønsberg
- Sweden (2):
  - Mölndal Hospital, Gothenburg
  - Universitety Hospital Örebro, Hudiksvall